CLINICAL TRIAL: NCT00652080
Title: An Open-Label Safety Study of API 31510 in a Topical Cream for in Situ Cutaneous Squamous Cell Carcinoma (SCCIS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BPGbio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTL0408
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Active Cream 3%; AM & PM
  Interventions: Drug: API 31510

INTERVENTIONS:
Drug: API 31510 — Topical Cream; 3% active; AM & PM application

SUMMARY:
The purpose of this study is to determine the safety and tolerability of pharmaceutical compound 31510 in a topical cream when applied to in situ cutaneous squamous cell carcinoma and to obtain preliminary efficacy data for the treatment of in situ cutaneous squamous cell carcinoma by Compound 31510 topical cream.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults > 18 years of age
* Primary, histologically confirmed SCCIS with a minimum area of 0.5 cm2 and with a maximum diameter of 2.0 cm target SCCIS lesion suitable for excision
* Histological diagnosis made no more than 4 weeks prior to the screening visit
* Histological biopsy removed 25% or less of the target lesion
* No other dermatological disease in the SCCIS target site or surrounding area
* Willing to refrain from using non-approved lotions or creams on the target site and surrounding area during the treatment period. Willing to refrain from washing the treated area for at least 8 hours following the application of study medication
* Willing to refrain from exposure to direct sunlight or ultraviolet light and to avoid the use of tanning parlors for the duration of the study
* Laboratory values for the tests listed in the Study Schedule on page 2 within the reference ranges as defined by the central laboratory, or "out of range" test results that are clinically acceptable to the investigator.
* Ability to follow study instructions and likely to complete all study requirements
* Written informed consent obtained, including consent for tissue to be examined and stored by the central dermatopathologist.
* Written consent to allow photographs of the target SCCIS lesion to be used as part of the study data
* For females of childbearing potential, a negative pregnancy test at screening and using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom, diaphragm, abstinence, or a monogamous relationship with a partner who has had a vasectomy)

Exclusion Criteria:

* Pregnant or lactating
* Presence of known or suspected systemic cancer
* Histological evidence of nBCC, sBCC, or any other tumor in the biopsy specimen
* Histological evidence of severe squamous metaplasia, infiltrative, desmoplastic or micronodular growth patterns in the biopsy specimen
* History of recurrence of the target SCCIS lesion
* Evidence of dermatological disease or confounding skin condition in the treatment area, e.g., BCC, actinic keratosis, rosacea, psoriasis, atopic dermatitis, eczema, xeroderma pigmentosa
* Concurrent disease or treatment that suppresses the immune system
* Chronic medical condition that in the judgment of the investigator(s) would interfere with the performance of the study or would place the patient at undue risk
* Known sensitivity to any of the ingredients in the study medication
* Use of a tanning parlor or other excessive or prolonged exposure to ultraviolet light or direct sunlight during the course of the study
* Treatment with systemic chemotherapeutic agents within the 6 months prior to the screening visit
* Use of systemic retinoids within the 6 months prior to the screening period
* Treatment with systemic immunomodulators or immunosuppressants within the 6 months prior to the screening period
* Use of topical immunomodulators within 2 cm of the target SCCIS lesion within the 4 weeks prior to the screening period
* Treatment with the following topical agents within the 4 weeks prior to the screening visit; levulinic acid, 5-fluorouracil, corticosteroids, retinoids, diclofenac, hyaluronic acid, imiquimod
* Undergone a facial resurfacing procedure, i.e., chemical peel, laser resurfacing, dermabrasion, within the 6 months prior to the screening visit, if the target SCCIS lesion is on the face
* Treatment with liquid nitrogen, surgical excision or curettage within 2cm of the target SCCIS lesion during the 4 weeks prior to the screening visit
* Elective surgery within 4 weeks prior to the screening visit, during the study, or 4 weeks after the treatment period
* Evidence of current chronic alcohol or drug abuse
* Current enrollment in an investigational drug or device or participation in such a study within 4 weeks of the screening visit
* In the investigator's opinion, evidence of unwillingness, or inability to follow the restrictions of the protocol and complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Burke Pharmaceuticals, Hot Springs, Arkansas
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Glazer Dermatology, Buffalo Grove, Illinois
  - Long Island Skin Cancer and Dermatalogic Surgery, PC, Smithtown, New York
  - Education and Research Foundation, Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were required to have at least one histologically-confirmed SCCIS lesion that was suitable for excision, ie, to have a lesion with a minimum area of 0.5 cm2 and a maximum diameter of 2.0 cm.
Groups:
- API 31510 Topical Cream: Active Cream 3%; AM & PM
  API 31510: Topical Cream; 3% active; AM & PM application
Period: Overall Study
Arm/Group | API 31510 Topical Cream
Started | 35
Completed | 31
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | API 31510 Topical Cream
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: To determine the safety and tolerability of API 31510 cream 3%, topically applied to in situ cutaneous squamous cell carcinomas (SCCIS).
Time Frame: 6 weeks
Population: Safety Population: All subjects who took at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Safety Population: Active Cream 3%; AM & PM
  API 31510: Topical Cream; 3% active; AM & PM application
Arm/Group | Safety Population
Number analyzed (Participants) | 35
Participants
  Subjects with an AE (Mild) | 10
  Subjects with an AE (Moderate) | 4
  Subjects with an AE (Severe) | 1
  Subjects without an AE | 20

2. Secondary Outcome: Percentage of Participants With a Complete Response
Description: To obtain a preliminary determination of the efficacy of API 31510 cream 3%,topically applied to in situ cutaneous squamous cell carcinomas.
  The subject was considered to have had a complete response only if the histological examination of the target lesion was negative.
Time Frame: 6 weeks
Population: Intent-to-Treat (ITT) Population: All subjects who were dispensed the study drug were included in this population.
  Per Protocol (PP) Population: All subjects who had SCCIS confirmed via histological results at baseline, had a Week 6 histological examination, and did not miss any interim visits.
Measure: Count of Participants; unit: Participants
Groups:
- ITT Population; PP Population: Active Cream 3%; AM & PM
  API 31510: Topical Cream; 3% active; AM & PM application
Arm/Group | ITT Population | PP Population
Number analyzed (Participants) | 34 | 27
Participants | 8 | 5

ADVERSE EVENTS:
Time Frame: All subjects in this study were treated with a formulation of CoQ10 3% topical cream that was applied twice daily for 6 weeks. The mean duration (SD) of treatment was 41.4 days (6.7) and ranged from 21 to 47 days.
Groups:
- 1 Safety Population: Active Cream 3%; AM & PM
  API 31510: Topical Cream; 3% active; AM & PM application
Arm/Group | 1 Safety Population
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 22/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Safety Population (N=35)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Safety Population (N=35)
Application site erythema (Skin and subcutaneous tissue disorders) | 7 (7)
Application site dryness (Skin and subcutaneous tissue disorders) | 1 (1)
Application site exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Application site bleeding (General disorders) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes